CLINICAL TRIAL: NCT01031563
Title: Risk Perception in Drug-Dependent Adults With and Without Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Maryland (Other)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909447; 09-DA-N447
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-05-03

CONDITIONS: Cocaine Dependence; Cannabis Dependence; Schizophrenia
Keywords: Risk Taking; Schizophrenia; Drug Abuse/Dependence; Comorbidity; Impulsivity; Drug Abuse
MeSH Terms: conditions — Cocaine-Related Disorders; Marijuana Abuse; Schizophrenia; Risk-Taking; Substance-Related Disorders; Impulsive Behavior

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

* Several studies of risk perception have demonstrated a common bias known as unrealistic optimism, in which individuals feel they are less likely than other people to experience unpleasant or harmful events in their lives, but more likely to experience pleasant or beneficial events.
* Previous research has indicated that individuals with schizophrenia have less of a sense of unrealistic optimism about adverse events than individuals without schizophrenia. However, research on risk perception in schizophrenia is sparse, primarily reporting on behaviors and decisions in the laboratory that likely are influenced by risk perception.
* Risk perception among substance users may be viewed in two separate categories: perception of vulnerability to adverse events and perception of vulnerability to negative outcomes associated with substance use. Research in both areas has yielded mixed results. Researchers are interested in studying the connections among schizophrenia, addiction, and risk perception in order to develop better drug use prevention and treatment programs for people with and without schizophrenia.

Objectives:

- To compare unrealistic optimism bias in people with and without schizophrenia and/or drug dependence, and its association with actual risky behavior.

Eligibility:

* Individuals between 18 and 64 years of age who fall into one of the following study categories:
* diagnoses of both drug dependence (marijuana or cocaine) and schizophrenia/schizoaffective disorder
* diagnosis of drug dependence only (marijuana or cocaine)
* diagnosis of schizophrenia/schizoaffective disorder only
* healthy volunteers with no history of drug use or serious mental disorder

Design:

* The study will require a single visit to the research center for a 5- to 6-hour session.
* Participants will complete questionnaires on medical and behavioral history, complete tests of thinking skills like memory and attention, complete a brief computerized decision-making task, and answer questions about risk perception.
* Participants will also provide urine samples and breath carbon monoxide measurements to test for recent use of tobacco and other substances.

DETAILED DESCRIPTION:
Background:

Several studies of risk perception have demonstrated a common bias known as unrealistic optimism', in which individuals feel they are less likely than other people to experience unpleasant or harmful events in their lives, but more likely to experience pleasant or beneficial events. In a previous study, we showed that unrealistic optimism about adverse events in patients with schizophrenia was lower than in healthy controls.

Objective:

To compare unrealistic optimism bias in people with and without schizophrenia and/or drug dependence, and its association with actual risky behavior.

Study Population:

Adults with current diagnosis (DSM-IV criteria) of schizophrenia or schizoaffective disorder (n = 24), with current drug dependence (cannabis or cocaine) (n = 24), with both schizophrenia and drug dependence (n = 24), or healthy, non-drug-using controls (n = 24).

Study Design:

Subjects will have a single study visit, at which their psychiatric and substance use histories, current substance use (urine drug testing, expired breath CO), risk perception, risk-taking/impulsivity, sensation-seeking, insight, history of risky behavior, and cognitive function will be assessed.

Outcome Measures:

Scores on Risk Perception Questionnaire, Balloon Analog Risk Task, short form self-report assessments of risk perception, risk-taking/impulsivity and sensation-seeking, Revised Life Orientation Scale, Self-Mastery Scale, Zuckerman-Kuhlman Personality Questionnaire, Repeatable Battery for the Assessment of Neuropsychological Status. South Oaks Gambling Screen-Revised, NORC DSM-IV Screen for Gambling Problems.

Benefit:

There is no direct benefit to subjects from study participation. Future benefits to society might be better understanding of risk perception biases associated with co-occurring substance abuse and schizophrenia, leading to development of more effective prevention and treatment programs and improved processes for obtaining informed consent.

Risks:

This study poses minimal risk to subjects, primarily boredom or anxiety from taking questionnaires and psychological tests and embarrassment from giving an observed urine specimen for drug testing.

ELIGIBILITY:
* Participants in three patient groups will have a current diagnosis of schizophrenia (or schizoaffective disorder), drug dependence, or both. Healthy comparison participants will be free of either diagnosis. Psychiatric diagnoses will be based on DSM-IV criteria as determined by the Structured Clinical Interview for DSM-IV (SCID; First et al 1997), which will be administered in either a computerized version or in the standard interview format. Participants in all four groups will be 18-64 years old, of either gender and of any race/ethnicity. Specific inclusion and exclusion criteria for the participant groups are as follows:

  1. Group 1: Drug dependence with schizophrenia or schizoaffective disorder

     Inclusion: Drug dependence; schizophrenia or schizoaffective disorder

     Exclusions: mood disorder; obsessive-compulsive disorder (OCD)
  2. Group 2: Drug dependence without schizophrenia or schizoaffective disorder

     Inclusion: Drug dependence.

     Exclusions: schizophrenia or schizoaffective disorder; mood disorder; OCD.
  3. Group 3: Schizophrenia or schizoaffective disorder without drug dependence

     Inclusion: DSM-IV schizophrenia or schizoaffective disorder.

     Exclusions: mood disorder; OCD; use of illegal drugs more than 3 times in the previous month.
  4. Group 4: Healthy comparison participants

     Exclusions: Any DSM-IV Axis I diagnosis (except simple phobia); use of illegal drugs more than 3 times in the previous month.
  5. Exclusions for all groups: History of neurological disease/condition (unrelated to schizophrenia or drug dependence) with ongoing cognitive sequelae; physical limitations (e.g., with hearing, vision or movement) that would prevent performance of computerized tasks; documented mental retardation.
  6. Substances of choice among drug-dependent participants (Groups 1 and 2) must be marijuana, cocaine or both (the commonest illegal drugs of abuse among patients with schizophrenia).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-08-18; Study Completion 2012-05-03

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- Maryland Psychiatric Research Center (MPRC) 55 Wade Avenue, Catonsville, Maryland, United States

REFERENCES:
- [Background] Marsch LA, Bickel WK, Badger GJ, Quesnel KJ. The anatomy of risk: a quantitative investigation into injection drug users' taxonomy of risk attitudes and perceptions. Exp Clin Psychopharmacol. 2007 Apr;15(2):195-203. doi: 10.1037/1064-1297.15.2.195. PMID 17469943
- [Background] Prentice KJ, Gold JM, Carpenter WT Jr. Optimistic bias in the perception of personal risk: patterns in schizophrenia. Am J Psychiatry. 2005 Mar;162(3):507-12. doi: 10.1176/appi.ajp.162.3.507. PMID 15741467
- [Background] Cherpitel CJ. Alcohol, injury, and risk-taking behavior: data from a national sample. Alcohol Clin Exp Res. 1993 Aug;17(4):762-6. doi: 10.1111/j.1530-0277.1993.tb00837.x. PMID 8214410